CLINICAL TRIAL: NCT05584579
Title: the Role of Laparoscopy in Lower Gastrointestinal Surgical Emergencies in Adults.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: zagazig 13
Record Dates: First submitted 2022-10-08; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Emergencies
Keywords: Emergency surgery; laparoscopy; lower abdominal surgery
MeSH Terms: conditions — Emergencies | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic surgery — laparoscopic surgery

SUMMARY:
Introduction: causes of lower abdominal pain caused by various GIT emergencies, including acute appendicitis, intestinal obstruction, acute perforated diverticulitis, obstructed hernia, and iatrogenic colon perforation. The role of Laparoscopy may be of diagnostic and therapeutic value.

Methods: Between April 2017 and April 2020, 793 patients were admitted to Zagazig University Hospital's emergency surgery unit with lower GIT emergencies, including acute appendicitis, acute intestine obstruction, complicated colonic diverticulum, complicated hernias, and iatrogenic colonic perforations.

DETAILED DESCRIPTION:
An acute lower abdomen is typically caused by peritoneal irritation caused by an abdominal organ's inflammation, rupture, or a hollow organ obstruction. Patients with severe acute lower abdominal pain either proceed to the operative room or additional investigations or diagnostic Laparoscopy (DL). Laparoscopy should not be used routinely for every acute lower abdomen case due to anesthetic risks and morbidity .

Most hospitals do emergency abdominal surgeries, and laparotomy in these procedures is associated with high death rates (14 to 20%) . Laparoscopic surgery has become a standard method for abdominal emergencies as a diagnostic and therapeutic tool. It has even been employed in some situations of lower abdominal crises in recent years .

The general surgeon frequently faces diagnostic challenges in emergency abdominal conditions. The diagnosis is crucial for planning the appropriate abdominal incision and avoiding unnecessary surgery. Noninvasive diagnostic approaches such as radiological examinations are not always conclusive. Furthermore, they are costly and cannot be performed 24 hours a day in all hospital circumstances . A retrospective observational study was designed to analyze the outcomes of a laparoscopic technique in emergent lower GIT surgeries regarding intraoperative and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old, both sexes, and have undergone laparoscopic surgery for acute lower GIT emergencies such as acute appendicitis, acute intestine obstruction, complicated colonic diverticulum, complicated hernias, and iatrogenic colonic perforations

Exclusion Criteria:

* less than 18 years of age and open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between April 2017 and April 2020, 793 patients were admitted to Zagazig University Hospital's emergency surgery unit with lower GIT emergencies, including acute appendicitis, acute intestine obstruction, complicated colonic diverticulum, complicated hernias, and iatrogenic colonic perforations. To be eligible for the study, patients must meet all of the following criteria: be >18 years old, both sexes, and have undergone laparoscopic surgery for acute lower GIT emergencies such as acute appendicitis, acute intestine obstruction, complicated colonic diverticulum, complicated hernias, and iatrogenic colonic perforations. The exclusion criteria were less than 18 years of age and open surgery. STROBE criteria were followed when reporting the work and registered in clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
intraoperative complications | up to 2 years

SECONDARY OUTCOMES:
postoperative complications | within 2 years of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No